CLINICAL TRIAL: NCT07388355
Title: WearLinq eWave Patch Study
Brief Title: A Usability Study of a Multi-channel ECG Monitoring Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wearlinq (Industry)
Collaborators: ABio Clinical Research Partners (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CLN 0001
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Participants; Heart Disease; Arrythmia; Cardiac
Keywords: Electrocardiogram; ECG; EKG; Cardiac diagnostic
MeSH Terms: conditions — Heart Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 7 Day Study (Experimental): Participants will receive and apply the WearLinq patch for 7 consecutive days
  Interventions: Device: eWave Patch
- Extended Use Cohort (Experimental): Participants will receive and apply the WearLinq patch for 30 consecutive days
  Interventions: Device: eWave Patch

INTERVENTIONS:
Device: eWave Patch — This device is a wearable multi-channel ECG monitoring device for continuous cardiac rhythm tracking.

SUMMARY:
This study it to evaluate the usability of the WearLinq eWave patch in a general adult population.

DETAILED DESCRIPTION:
Once eligibility is determined, participants will receive and apply the WearLinq patch for 7 consecutive days (or until an endpoint is met). A subset of subjects will be asked to participate in an Extended Use Cohort (30 days).

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old and able to consent
* Capable of using a smartphone app
* Willing to shave patch area if needed

Exclusion Criteria:

* Planning to undergo an MRI during the study period
* Known allergic reaction to adhesives or hydrogels or with family history of adhesive skin allergies, or any other dermatological conditional that could confound placement or results
* Presence of pacemaker, ICD or other implanted electronic devices
* Open wounds, lesions or infected or inflamed areas of skin at the placement site (left-center of chest/sternum)
* Pregnant or intending to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Wear Duration | 7 Days
  Days of use until one of the following is reached: patch no longer adheres, signal loss, voluntary removal, or 7 days is achieved
Adverse Events | 7 Days
  Incidences of self-reported adverse events for the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Chris Daniel, Study Director — WearLinq, Inc.
Locations (1):
- ABio Clinical Research Partners, New London, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No plans to be provided/Not applicable